CLINICAL TRIAL: NCT03259061
Title: A Study of Border Line Cases of Velopharyngeal Incompetence and Insufficiency Using Cephalometry and Nasofibroscopy
Brief Title: A Study of Border Line Cases of Velopharyngeal Incompetence Using Cephalometry and Nasofibroscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AbdElAzeez Mohammad Faheem Darweesh, Dr, Assiut University
Other Study IDs: Border line VPI study
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Velopharyngeal Insufficiency
MeSH Terms: conditions — Velopharyngeal Insufficiency | interventions — Cephalometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Flexible fiberoptic nasopharyngoscopy — 1. Flexible fiberoptic nasopharyngoscopy (FFN) allows direct transnasal observation of the anatomy and dynamic activity of the velopharyngeal sphincter. Such observations can be recorded for permanent documentation by coupling FFN to a video camera with simultaneous audio recording. Numerous published reports discuss the advantages of FFN as a clinical method for evaluating velopharyngeal function during speech (10).
  2. Cephalometric analysis, is the clinical application of cephalometry. It is analysis of the dental and skeletal relationships of a human skull and is frequently used by dentists, orthodontists, and oral and maxillofacial surgeons as a treatment planning tool.
  Cephalometric analysis can also be applied for assessing the velopharyngeal structure and function. More specifically, velopharyngeal function in terms of its shape and mobility was analyzed quantitatively on the basis of cephalometric principle
  Other Names: Cephalometry

SUMMARY:
The aim of this work is to evaluate the role of cephalometry &nasofibroscopy as objective tools in order to confirm the diagnosis based upon the clinical judgment of border line cases suspected to have velopharyngeal incompetence or insufficiency.

DETAILED DESCRIPTION:
The velopharyngeal mechanism is constituted by the muscles of the soft palate, posterior and lateral pharyngeal walls (1), separating the oropharynx from the nasopharynx. Such structures, particularly the soft palate, play a key role in the velopharyngeal closure physiology (2). Velopharyngeal closure patterns may be classified as follows: coronal, where there is predominant soft palate movement toward the posterior pharyngeal wall; sagittal, where there is predominant movement of the lateral pharyngeal walls toward the pharynx midline; circular, where balanced movements of lateral pharyngeal walls and soft palate are observed; circular with Passavant's ridge, where the circular closure is associated with the development of a mucosal fold named Passavant's ridge on the posterior pharyngeal wall(3). The velopharyngeal closure allows the separation between the nasal and oral cavities during activities such as oral sounds emission, blowing, whistling, swallowing, sucking and vomiting reflex, respecting the level of closure demanded by each activity (4,5).

In cases where the structures of the velopharyngeal mechanism do not work properly, the presence of a space called velopharyngeal aperture is observed between them, characterizing a velopharyngeal dysfunction. One of the reasons for the occurrence of such an aperture is the shortage of soft palate tissue. This dysfunction is called velopharyngeal insufficiency and may be corrected either surgically or by prosthetic management followed by speech therapy. In cases where such dysfunction occurs because of a failure in the velopharyngeal structures movement, physiological or neuromotor deficiency, it is called velopharyngeal incompetence that may be eliminated by means of speech therapy (2,6). On the other hand, if such condition is a result of the presence of compensatory articulations or other speech learning errors, it does not reflect physical or neuromuscular alterations, constituting indication for speech therapy(7). Individuals with velopharyngeal dysfunction present hypernasality, nasal air emission, poor intraoral pressure, and may present associated nasal/facial movements and compensatory articulations during the emission of oral consonants (8,9).

Assessment of the velopharyngeal function can be done by the following procedures:

1. Flexible fiberoptic nasopharyngoscopy (FFN) allows direct transnasal observation of the anatomy and dynamic activity of the velopharyngeal sphincter. Such observations can be recorded for permanent documentation by coupling FFN to a video camera with simultaneous audio recording. Numerous published reports discuss the advantages of FFN as a clinical method for evaluating velopharyngeal function during speech (10).

   Flexible fiberoptic nasopharyngoscopy (FFN) is a valuable tool for direct visualization because it allows observation of the velopharyngeal valve during dynamic activity for a prolonged period with (1) Minimal interference of the structures involved and (2) No radiation exposure. Whereas most clinicians acknowledge the theoretic advantages of FFN and accept it as a valid technique for assessing velopharyngeal function, there are few published studies that have addressed the validity and reliability of endoscopic procedures (10). Endoscopic evaluation has high face validity, and several reports have indicated that FFN has good construct validity when compared with radiologic assessments (11).
2. Cephalometric analysis, is the clinical application of cephalometry. It is analysis of the dental and skeletal relationships of a human skull and is frequently used by dentists, orthodontists, and oral and maxillofacial surgeons as a treatment planning tool.

Cephalometric analysis can also be applied for assessing the velopharyngeal structure and function. More specifically, velopharyngeal function in terms of its shape and mobility was analyzed quantitatively on the basis of cephalometric principle (12,13).

Border line cases of velopharyngeal incompetence of insufficiency are known to be problematic and usually causes confusion for phoniatricians especially in patients who will undergo adenotonsillectomy. For this purpose, objective assessment is necessary to support or reject the clinical findings of VPI cases.

ELIGIBILITY:
Inclusion Criteria:

Patients must have border line velopharyngeal abnormality which was diagnosed clinically.

Ability to understand and the willingness to sign a written informed consent(if he was a child so his parents or his guardian should has tis ability)

Exclusion Criteria:

1. Mental Retardation.
2. Presence of Neurological deficit affecting speech.
3. Palatal paralysis or paresis.
4. Overt cleft palate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Comparison between Cephalometric and nasofibroscopic findings and clinical findings | Baseline
  Assessment of the function of velopharyngeal valve by nasofibroscopy and cephalometric measurements in clinically border line cases of velopharyngeal incompetence in order to ensure the presence of Velophayngeal incompetence

REFERENCES:
- [Background] Camargo LO, Rodrigues CM, Avelar JA. Oclusão velofaríngea em indivíduos submetidos à nasoendoscopia na Clínica de Educação para Saúde (CEPS) 20(1):35-48, 2001.
- [Background] Skolnick ML, McCALL GN, Barnes M. The sphincteric mechanism of velopharyngeal closure. Cleft Palate J. 1973 Jul;10:286-305. No abstract available. PMID 4513919
- [Background] Penido FA, Noronha RM, Caetano KI, Jesus MS, Di Ninno CQ, Britto AT. Correlação entre os achados do teste de emissão de ar nasal e da nasofaringoscopia em pacientes com fissura labiopalatina operada. Rev Soc Bras Fonoaudiol. 2007;12(2):126-34.
- [Background] Mourão D, Souza GS, Torres LV, Vaz RN, Prado SG. Estudo sobre desenvolvimento fonológico em fissurados: implicações na fala e na linguagem. Estudos. 2006;33(5/6):425-41.
- [Background] De Bodt M, Van Lierde K. Cleft palate speech and velopharyngeal dysfunction: the approach of the speech therapist. B-ENT. 2006;2 Suppl 4:63-70. PMID 17366850
- [Background] Trindade IE, Genaro KF, Yamashita RP, Miguel HC, Fukushiro AP. [Proposal for velopharyngeal function rating in a speech perceptual assessment]. Pro Fono. 2005 May-Aug;17(2):259-62. doi: 10.1590/s0104-56872005000200015. Portuguese. PMID 16909536
- [Background] Witt PD. Management of velopharyngeal dysfunction. In: Persing JA, Evans GR. Soft-tissue surgery of the craniofacial region. New York: Informa; 2007. p.113-28.
- [Background] Smith BE, Kuehn DP. Speech evaluation of velopharyngeal dysfunction. J Craniofac Surg. 2007 Mar;18(2):251-61; quiz 266-7. doi: 10.1097/SCS.0b013e31803ecf3b. PMID 17414269
- [Background] D'Antonio LL, Marsh JL, Province MA, Muntz HR, Phillips CJ. Reliability of flexible fiberoptic nasopharyngoscopy for evaluation of velopharyngeal function in a clinical population. Cleft Palate J. 1989 Jul;26(3):217-25; discussion 225. PMID 2758674
- [Background] Mourino AP, Weinberg B. A cephalometric study of velar stretch in 8 and 10-year old children. Cleft Palate J. 1975 Oct;12:417-35. PMID 1058753
- [Background] Simpson RK, Colton J. A cephalometric study of velar stretch in adolescent subjects. Cleft Palate J. 1980 Jan;17(1):40-7. PMID 6928116